CLINICAL TRIAL: NCT06452589
Title: A Pre-Market, First-In-Human, Pilot, Interventional, Clinical Investigation to Evaluate Safety and Feasibility of the FieldForce™ Ablation System in Patients With Atrial Fibrillation
Brief Title: The Field PULSE Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Field Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLN-PULSE-PR-01
Record Dates: First submitted 2024-06-05; First posted 2024-06-11 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Atrial Arrhythmias
Keywords: atrial arrhythmia; atrial fibrillation; PFA; Pulse Field Ablation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Irreversible Electroporation Therapy

STUDY DESIGN:
Intervention Model Description: Prospective single arm safety and feasibility study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Catheter ablation (Experimental): Adult patients with a history of atrial fibrillation or associated atrial arrhythmias and indicated for a catheter ablation.
  Interventions: Device: FieldForce Ablation System

INTERVENTIONS:
Device: FieldForce Ablation System — The FieldForce Ablation System is indicated for cardiac electrophysiologic mapping, delivery of diagnostic pacing stimuli, and pulse field ablation of cardiac tissue. When used with the FieldForce Ablation Catheter, the FieldForce System is intended to be used in the right/left atria and/or left/right ventricle to deliver PFA ablation lesions in the selected areas of the chamber.
  Other Names: Pulse Field Ablation

SUMMARY:
This is a pre-market, first-in-human, pilot, interventional, clinical investigation that aims to evaluate safety and feasibility of the FieldForce™ Ablation system in patients with atrial fibrillation who are indicated for an AF catheter ablation.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is a cardiac rhythm disorder characterized by irregular and often abnormally fast contractions of the atrial cardiomyocytes resulting in various symptoms, including palpitations, dizziness, shortness of breath and tiredness.

AF is the most common sustained cardiac arrhythmia, having a prevalence of about ≈2% in the general population. AF can be associated with increased morbidity and mortality in patients with cardiovascular disease, and increased risk of stroke in general population.

Catheter ablation for the treatment of AF is primarily performed with radiofrequency (RF) or cryoballoon (CB) catheters to achieve anatomic pulmonary vein isolation (PVI). However, the technical challenges of achieving effective PVI and recognized risks of complications are two most important factors driving the need for replacing thermal ablation technologies like RF and CB.

Pulsed field ablation (PFA) is a non-thermal ablation technology which uses high voltage pulsed electrical fields to ablate tissues. This destabilizes cell membranes by forming irreversible nanoscale pores and leakage of cell contents, culminating in cell death. Several clinical studies have demonstrated that PFA can achieve pulmonary vein isolation with minimal collateral damage in a time-efficient manner.

The FieldForce™ Ablation System utilizes PFA with an innovative electrode technology called FieldBending™ designed to improve safety, tolerability, and efficacy for focal deflectable catheters used for the treatment of AF.

ELIGIBILITY:
Inclusion Criteria:

1. Signed patient informed consent form (ICF).
2. Female and male patients aged ≥ 18 and ≤ 80.
3. Documented atrial fibrillation via an electrocardiogram (must be at least 30 seconds) within one year of enrollment.
4. Indicated for a first-time catheter ablation for atrial fibrillation or associated atrial arrhythmias (European guidelines).

Exclusion Criteria:

1. Body Mass Index > 40.
2. Ineligible for ablation (including but not limited to known left atrial thrombus).
3. AF secondary to electrolyte imbalance, thyroid disease, alcohol abuse or other reversible/non-cardiac causes.
4. Previous endocardial/epicardial ablation or surgery for AF.
5. NYHA Class IV.
6. Left atrial appendage device or occlusion within 180 days.
7. Atrial or ventricular septal defect closure.
8. Atrial myxoma.
9. The presence of inferior vena cava embolic protection filter devices.
10. Significant or symptomatic untreated hypotension, bradycardia, or chronotropic incompetence.
11. History of hemodynamically severe valvular disease. Severity should be assessed using echocardiography, according to AHA and European guidelines.
12. Diagnosis of pacemaker dependance.
13. Uncontrolled abnormal bleeding and/or clotting disorder.
14. Contraindication to systemic or oral anticoagulation.
15. Serious or untreated medical conditions that would prevent participation in the study, interfere with assessment of therapy, or confound data or its interpretation, including but not limited to solid organ or hematologic transplant, or currently being evaluated for an organ transplant.
16. History of severe lung disease, pulmonary hypertension, or any lung disease involving abnormal blood gases or significant dyspnea which may interfere with the assessment of the therapy.
17. Active malignancy.
18. Uncontrolled clinically significant infection.
19. Life expectancy is less than one year.
20. Clinically significant psychological condition that in the investigator's opinion would prohibit the subject's ability to meet the study requirements.
21. Any of the following within 3 months of enrollment: myocardial infarction, unstable angina, percutaneous coronary intervention, heart surgery (coronary artery bypass grafting/atriotomy), stroke or transient ischemic attack (TIA);
22. Participation in another investigational study that would interfere with this study.
23. Patient is not able to understand the nature of this study or is unwilling or unable to attend the study procedures.
24. Women who are of childbearing age and not on a reliable form of birth control.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-07-25 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of early and late onset adverse events | 30 days and 12 months
  Adverse events to evaluate the safety of the FieldForce™ Ablation System will be collected. The incidence of the major safety events will be evaluated.
Performance | index procedure and 3 months
  To characterize the proportion of subjects who achieved pulmonary vein isolation (PVI) using the FieldForce™ Ablation System

SECONDARY OUTCOMES:
Device or Procedure Related SAEs | 30 days, 3 months, 6 months and 12 months
  Proportion of subjects reporting one or more device-or procedure-related SAEs.
Presence of Atrial Arrhythmias from index procedure through end of study | 6 months and 12 months
  To evaluate freedom from atrial arrhythmia (including atrial fibrillation, flutter, or tachycardia).
Procedure Time | Index procedure
  To characterize procedure times (including total duration, transpired ablation time, fluoroscopy time).

CONTACTS AND LOCATIONS:
Locations (1):
- Na Homolce Hospital, Prague, Czechia